CLINICAL TRIAL: NCT04898010
Title: Investigator Initiated Pilot Study to Assess the Safety and Efficacy of a Selective Cytopheretic Device (SCD) to Treat ICU Patients With Acute Kidney Injury (AKI) and Hepatorenal Syndrome (HRS) Type I
Brief Title: The Selective Cytopheretic Device (SCD) for Acute Kidney Injury (AKI) and Hepatorenal Syndrome (HRS) Type I
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: On hold while seeking funding.
Sponsor: Lenar Yessayan (Other)
Responsible Party: Sponsor-Investigator, Lenar Yessayan, Associate Professor of Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00163117
Record Dates: First submitted 2021-05-18; First posted 2021-05-24 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Acute Kidney Injury; Hepatorenal Syndrome
MeSH Terms: conditions — Acute Kidney Injury; Hepatorenal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Selective Cytopheretic Device (Experimental): Subjects will be placed on Selective Cytopheretic Device (SCD) for planned daily 24 hour therapy for up to 7 consecutive days.
  Interventions: Device: Selective Cytopheretic Device

INTERVENTIONS:
Device: Selective Cytopheretic Device — The Selective Cytopheretic Device (SCD) treatment will be delivered using a two-cartridge system using a type of dialysis equipment commonly used for conventional hemodialysis therapy. The SCD cartridge will be added immediately post-hemofilter to the circuit of a standard hemodialysis system, and treatment will be delivered for 24 hours. Blood exchange will occur using a dialysis catheter.

SUMMARY:
This research study is being done to learn what effect 7 days of treatment with the Selective Cytopheretic Device (SCD) will have on these white blood cells in the bloodstream of patients with hepatorenal syndrome and to learn whether it has any effect on the blood circulation and kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis with ascites.
* Not currently listed for liver transplant.
* Worsening renal failure most likely due to Hepatorenal Syndrome Type I with low glomerular filtration rate (GFR).
* No sustained improvement in renal function after diuretic withdrawal and expansion of plasma volume with 1.5 liters of plasma expander.
* No sustained improvement in renal function or intolerant to treatment with octreotide and /or midodrine.
* Able to tolerate regional citrate anticoagulation and continuous renal replacement therapy (CRRT) for 24 hours or greater.
* Intent to deliver full supportive care through aggressive management utilizing all available therapies for a minimum of 96 hours.
* Receiving medical care in an intensive care unit.
* Absence of shock, ongoing bacterial infection and fluid losses, and current treatment with nephrotoxic medications, hepatocellular carcinoma.
* Females of child bearing potential who are not pregnant (confirmed by a negative serum pregnancy test) and not lactating if recently post-partum.
* Two (2) consecutive intra-circuit Ionized Calcium (iCa) levels <0.40 Millimoles per liter (mmol/L), at least 30 minutes apart.

Exclusion Criteria:

* Evidence of chronic kidney disease Stage 4.
* Patients with Model for End-Stage Liver Disease (MELD) score > 40 (since these patients are unlikely to survive a 90-day follow-up period).
* Acute or chronic use of circulatory support device.
* Mechanical ventilation for greater than 7 consecutive days.
* AKI occurring in the setting of burns, obstructive uropathy, allergic interstitial nephritis, acute or rapidly progressive glomerulonephritis, vasculitis, hemolytic uremic syndrome, thrombotic thrombocytopenic purpura (TTP), malignant hypertension, scleroderma renal crisis, atheroembolism, functional or surgical nephrectomy, cyclosporine or tacrolimus nephrotoxicity. No evidence of intrinsic parenchymal renal disorder, ultrasonic evidence of obstructive uropathy or proteinuria greater than 500 mg/day.
* Presence of any organ transplant at any time.
* Metastatic malignancy which is actively being treated or may be treated by chemotherapy or radiation during the subsequent three-month period after study protocol therapy.
* Severe, uncontrolled cardiac disease.
* Chronic immunosuppression.
* Medical history of HIV or AIDS.
* Current Do Not Attempt Resuscitation (DNAR), Allow Natural Death (AND), or withdrawal of care status, or anticipated change in status within the next 7 days.
* Patient is moribund or chronically debilitated for whom full supportive care is not indicated.
* Dry weight >150 kg.
* Platelet count <30,000/mm3.
* Concurrent enrollment in another interventional clinical trial. Patients enrolled in clinical studies where only measurements and/or samples are taken (i.e., no test device or test drug used) are allowed to participate
* Use of any other investigational drug or device within the previous 30 days
* Patient is a prisoner.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of serious adverse events related to selective cytopheretic device (SCD) | Up to 90 days
Number of deaths related to selective cytopheretic device | Up to 90 days
Number of events of significant clotting within the device as assessed by visual inspection | Up to 7 days
  Source documentation will record either present, absent, or not-assessed
Number of unforeseen malfunction(s) that results in the need for discontinuation | Up to 7 days
Number if events with evidence of leakage (i.e., cracking/breakage of a port, connector, SCD casing cartridge or tubing). | Up to 7 days

SECONDARY OUTCOMES:
Dialysis independence | Up to 90 (+/- 7 days)
  Dialysis independence at days 1-5 post SCD, and at days 30 and 90 (+/- 7 days). Dialysis independence will be assessed using the medical record.
Change in renal function | Baseline (prior to dialysis), days 1-5 post SCD, days 30 and 90 (among survivors and those free from dialysis) (+/- 7 days)
  As measured by serum creatinine from baseline (prior to dialysis initiation) at days 1-5 post SCD and at days 30 and 90 (among survivors and those free from dialysis).
Change in liver function | Baseline, at days 1-5 post SCD or until ICU discharge (if earlier than 5 days) and at days 30 and 90 (among survivors)
  Measured by blood tests of liver function parameters such as AST, ALT, alkaline phosphatase
Change in liver function | Baseline (prior to dialysis), Days 1-5 post SCD or until ICU discharge (if earlier than 5 days) and at days 30 and 90 (among survivors) (+/- 7 days).
  Measured by blood test of bilirubin
Change in coagulation parameters | Baseline (prior to dialysis), Days 1-5 post SCD or until ICU discharge (if earlier than 5 days) and at days 30 and 90 (among survivors) (+/- 7 days).
  Coagulation parameters include Prothrombin Time (PT), Activated Partial Thromboplastin Time (PTT), and International Normalized Ratio (INR) all reported in seconds
Change in model for end-stage liver disease (MELD) score | Baseline (prior to dialysis), Days 1-5 post SCD or until ICU discharge (if earlier than 5 days) and at days 30 and 90 (among survivors) (+/- 7 days).
  MELD score is a number that ranges from 6 (least sick) to 40 (most sick) based on blood tests which ranks the degree of sickness from liver disease.

CONTACTS AND LOCATIONS:
Overall Officials: Lenar Yessayan, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yessayan LT, Sharma P, Westover AJ, Szamosfalvi B, Humes HD. Extracorporeal Immunomodulation Therapy in Acute Chronic Liver Failure With Multiorgan Failure: First in Human Use. ASAIO J. 2024 Mar 1;70(3):e53-e56. doi: 10.1097/MAT.0000000000002033. Epub 2023 Aug 29. PMID 37643314